CLINICAL TRIAL: NCT05148780
Title: Acute Respiratory Infections Global Outpatient Study
Brief Title: A Study of Acute Respiratory Infections in Global Outpatient Setting
Acronym: ARGOS
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CR109104; NOPRODRSV4002 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2021-11-25; First posted 2021-12-08 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Acute Respiratory Infection
Keywords: Respiratory syncytial virus (RSV); Flu; COVID-19
MeSH Terms: conditions — Influenza, Human; COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Participants with Acute Respiratory Infections (ARI) in Outpatient Setting (Other): Participants presenting with ARIs in an outpatient setting who are at high risk of progressing to severe disease will be screened for viral respiratory pathogens (respiratory syncytial virus [RSV], Influenza, severe acute respiratory syndrome coronavirus 2 [SARS-COV-2]) by collecting a nasal swab. If a participant is positive for RSV and/or influenza virus and/or SARS-CoV-2 based on a study test or standard-of-care (SOC) polymerase chain reaction (PCR)-based test, the participant will be eligible for enrollment in the study in the home-based short-term and long-term follow-up phases.
  Interventions: Diagnostic Test: Nasal Swab Sample

INTERVENTIONS:
Diagnostic Test: Nasal Swab Sample — Nasal swab sample will be used to screen participants for detection of viral pathogens. No intervention or study drug will be administered as part of this study.

SUMMARY:
The purpose of this study is to evaluate the positivity rate of respiratory syncytial virus (RSV), influenza virus and severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) in high-risk participants presenting with acute respiratory infections (ARIs) in outpatient settings during the influenza/RSV season and to evaluate the association between lower respiratory tract disease (LRTD) and ARI-related hospitalization in participants positive for RSV.

DETAILED DESCRIPTION:
Lower respiratory tract infections (LRTIs) are a major cause of mortality and morbidity worldwide with 2.3 million deaths in 2016 alone among all age groups, making it the sixth leading cause of mortality. The current study aims to assess the burden of RSV infections among adult participants presenting in outpatient settings, who are at high risk of complications or progression to severe disease due to their age or pre-existing comorbidities. Regional data from the United States (US), Europe, Middle East, and Asia (EMEA) and Asia-Pacific (APAC) will provide evidence on local RSV morbidity, mortality, medical resource utilization (MRU), standard of care, and quality of life in adults participants. A subset of participants positive for influenza virus and/or SARS-CoV-2 will also be enrolled, to allow for a comparative assessment of disease burden between the 3 viral respiratory pathogens. No study drug will be involved in this study. The total duration of the study for each participant will be a maximum of 3 months (+-1 week) from the date of enrollment. Safety will be assessed in the form of adverse events and serious adverse events related to study devices or procedures and for deaths regardless of causality.

ELIGIBILITY:
Inclusion Criteria:

* Present to the general physician (GP)/specialist outpatient settings/respiratory clinics or in Emergency department (ED) settings with symptoms suggestive of a diagnosis of Acute Respiratory Infections (ARI)
* For inclusion in the home-based follow-up phases, must test positive for respiratory syncytial virus (RSV) and/or influenza and/or Severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) per a molecular-based diagnostic assay (polymerase chain reaction [PCR]-based) using a nasal swab (nasopharyngeal or similar) sample. Co-infections are permitted to be enrolled in the study
* Must be able to read, understand, and complete questionnaires
* Must be willing to provide verifiable identification, has means to be contacted and to contact the investigator during the study
* Willing and able to adhere to the specifications in this protocol

Exclusion Criteria:

* Has a clinical condition other than those as specified in study protocol which, in the opinion of the investigator, could prevent, confound, or limit the protocol-specified assessments
* Received an investigational drug (including investigational vaccines) within 3 months before the start of the study or the first data collection time-point
* Is currently enrolled or plans to participate in another investigational study on RSV, influenza or SARS-CoV-2 during the current study
* Is, in the opinion of the investigator, unlikely to adhere to the requirements of the study, or is unlikely to complete the full course of observation
* Cannot communicate reliably with the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 245 (Actual)
Dates: Start 2021-12-20 (Actual); Primary Completion 2023-02-20 (Actual); Study Completion 2023-02-22 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants Positive for Respiratory Syncytial Virus (RSV) | Day 1
  Percentage of participants positive for RSV, among those screened for viral pathogens using a polymerase chain reaction (PCR)-based test will be reported.
Percentage of Participants Positive for Influenza Virus | Day 1
  Percentage of participants positive for influenza virus, among those screened for viral pathogens using a PCR-based test will be reported.
Percentage of Participants Positive for Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2) | Day 1
  Percentage of participants positive for SARS-CoV-2, among those screened for viral pathogens using a PCR- based test will be reported
Number of Participants with Relative Risk of Acute Respiratory Infections (ARI)- related Hospitalization in Participants Positive for RSV with Lower Respiratory Tract Disease (LRTD) or Without LRTD | Up to 3 months
  Number of participants with relative risk of ARI-related hospitalization in participants positive for RSV with LRTD or without LRTD will be reported. LRTD is defined as new onset or worsening from chronic condition of 3 or more of the below symptoms as captured in the Respiratory Infection Intensity and Impact Questionnaire (RiiQTM) V2 at the same assessment time-point: Cough, Short of breath, Coughing up phlegm (sputum), Wheezing.

SECONDARY OUTCOMES:
Number of Participants with Relative Risk of ARI-related Hospitalization in Participants Positive for Influenza Virus Diagnosed with or Without LRTD | Up to 3 months
  Number of participants with relative risk of ARI-related hospitalization in participants positive for influenza virus diagnosed with or without LRTD will be reported. LRTD is defined as new onset or worsening from chronic condition of 3 or more of the below symptoms as captured in the RiiQTM V2 at the same assessment time-point: Cough, Short of breath, Coughing up phlegm (sputum), Wheezing.
Number of Participants with Relative Risk of ARI-related Hospitalization in Participants Positive for SARS-CoV-2 with or Without LRTD | Up to 3 months
  Number of participants with relative risk of ARI-related hospitalization in participants positive for SARS-CoV-2 with or without LRTD will be reported. LRTD is defined as new onset or worsening from chronic condition of 3 or more of the below symptoms as captured in the RiiQTM V2 at the same assessment time-point: Cough, Short of breath, Coughing up phlegm (sputum), Wheezing
Percentage of Participants Positive for RSV Reporting ARI-related Hospitalizations During the Study Period | Up to 3 months
  Percentage of participants positive for RSV reporting ARI-related hospitalizations during the study period will be reported.
Percentage of Participants Positive for Influenza Virus Reporting ARI-related Hospitalizations During the Study Period | Up to 3 months
  Percentage of participants positive for influenza virus reporting ARI-related hospitalizations during the study period will be reported.
Percentage of Participants Positive for SARS-CoV-2 Reporting ARI-related Hospitalizations During the Study Period | Up to 3 months
  Percentage of participants positive for SARS-CoV-2 reporting ARI-related hospitalizations during the study period will be reported.
Time to ARI- related Hospitalization in Participants Positive for RSV | Up to 3 months
  Time to ARI- related hospitalization in participants positive for RSV will be reported.
Time to ARI- related Hospitalization in Participants Positive for Influenza Virus | Up to 3 months
  Time to ARI- related hospitalization in participants positive for influenza virus will be reported.
Time to ARI- related Hospitalization in Participants Positive for SARS-CoV-2 | Up to 3 months
  Time to ARI- related hospitalization in participants positive for SARS-CoV-2 will be reported.
Percentage of Participants Presenting with Complications at Screening and Diagnosed with or Without LRTD | Day 1
  Percentage of participants presenting with complications at screening and diagnosed with or without LRTD will be reported.
Percentage of Participants Reporting ARI- related Complications During the Follow-up Period and Diagnosed with or Without LRTD | Up to 3 months
  Percentage of participants reporting ARI- related complications during the follow-up period and diagnosed with or without LRTD will be reported.
Time to ARI- related Complications During the Follow-up Period in Participants Positive for RSV | Up to 3 months
  Time to ARI- related complications during the follow-up period in participants positive for RSV will be reported.
Time to ARI- related Complications During the Follow-up Period in Participants Positive for Influenza Virus | Up to 3 months
  Time to ARI- related complications during the follow-up period in participants positive for influenza virus will be reported.
Time to ARI- related Complications During the Follow-up Period in Participants Positive for SARS-CoV-2 | Up to 3 months
  Time to ARI- related complications during the follow-up period in participants positive for SARS-CoV-2 will be reported
Percentage of Participants Presenting with Clinically Relevant Disease at Screening and Diagnosed with or Without LRTD | Day 1
  Percentage of participants presenting with clinically relevant disease at screening and diagnosed with or without LRTD will be reported.
Percentage of Participants Reporting ARI- related Clinically Relevant Disease During the Follow-up Period and Diagnosed with or Without LRTD | Up to 3 months
  Percentage of participants reporting ARI-related clinically relevant disease during the follow-up period and diagnosed with or without LRTD will be reported.
Time to ARI-related Clinically Relevant Disease During the Follow-up Period in Participants Positive for RSV | Up to 3 months
  Time to ARI-related clinically relevant disease during the follow-up period in participants positive for RSV will be reported.
Time to ARI-related Clinically Relevant Disease During the Follow-up Period in Participants Positive for Influenza Virus | Up to 3 months
  Time to ARI-related clinically relevant disease during the follow-up period in participants positive for influenza virus will be reported.
Time to ARI-related Clinically Relevant Disease During the Follow-up Period in Participants Positive for SARS-CoV-2 | Up to 3 months
  Time to ARI-related clinically relevant disease during the follow-up period in participants positive for SARS-CoV-2 will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (72):
- United States (39):
  - Central Alabama Research, Birmingham, Alabama
  - Lakeview Clinical Research, Guntersville, Alabama
  - Synexus Clinical Research US Inc, Mesa, Arizona
  - Fiel Family and Sports Medicine Clinical Research Advantage, Phoenix, Arizona
  - Harrisburg Family Medical Center, Harrisburg, Arkansas
  - Innovative Research of West Florida, Incorporated, Clearwater, Florida
  - New Life Medical Research Center, Inc., Hialeah, Florida
  - Best Quality Research Inc, Hialeah, Florida
  - PharmaDUX Clinical Medical Research, LLC, Medley, Florida
  - Homestead Associates in Research,Inc, Miami, Florida
  - Alma Clinical Research, Miami, Florida
  - Research Institute of South Florida Inc, Miami, Florida
  - Pines Care Research Center Inc, Pembroke Pines, Florida
  - Santos Research Center, Tampa, Florida
  - Columbus Regional Research Institute, Columbus, Georgia
  - IACT Health, Rincon, Georgia
  - Snake River Research, PLLC, Idaho Falls, Idaho
  - Washington University School Of Medicine, St Louis, Missouri
  - Montana Medical Research, Missoula, Montana
  - Healor Primary Care, Las Vegas, Nevada
  - Las Vegas Medical Research, Las Vegas, Nevada
  - Santa Rosa Medical Centers of Nevada, Las Vegas, Nevada
  - Urgent Care Clinical Trials at AFC Urgent Care, The Bronx, New York
  - Montefiore Medical Center, The Bronx, New York
  - American Health Network, LLC, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - DayStar Clinical Research, Inc., Akron, Ohio
  - Urgent Care Clinical Trials at AFC Urgent Care, Easley, South Carolina
  - Premier Family Physicians, Carrollton, Texas
  - Next Level Urgent Care, Corpus Christi, Texas
  - Southwest Family Medicine Associates, Dallas, Texas
  - Urgent Care Clinical Trials Fort Worth, Fort Worth, Texas
  - Southwest Clinical Trials, Houston, Texas
  - Renovatio Clinical, Magnolia, Texas
  - Benchmark Research, San Angelo, Texas
  - CCT Research at Olympus Family Medicine, Holladay, Utah
  - CCT Research at South Ogden Family Medicine, Ogden, Utah
  - Clinical Research Partners, LLC, Henrico, Virginia
  - IACT Health, Suffolk, Virginia
- ALTA Clinical Research Inc., Edmonton, Alberta, Canada
- France (3):
  - CHU Grenoble, La Tronche
  - Hopital Edouard Herriot - CHU Lyon, Lyon
  - CHU Nimes Hopital Caremeau, Nîmes
- Japan (3):
  - Fujita Health University Hospital, Date-gun
  - Hanasaki Clinic, Kiyosu-shi
  - Miyagikoseikyokai Saka General Hospital, Shiogama
- Malaysia (4):
  - Klinik Kesihatan Putrajaya Presint 9, Kuala Lumpur
  - Klinik Kesihatan Kuang, Kuang
  - Klinik Kesihatan Masjid Tanah, Masjid Tanah
  - Hospital Miri, Miri
- Poland (5):
  - Gabinet Lekarski Pediatryczno-Alergologiczny, Bialystok
  - NEURO MEDIC Janusz Zbrojkiewicz Poradnia Wielospecjalistyczna, Katowice
  - ETG Lodz, Lodz
  - EMC Instytut Medyczny SA PL CERTUS, Poznan
  - NZOZ Leczniczo Rehabilitacyjny Osrodek Medycyny Rodzinnej, Wroclaw
- South Korea (4):
  - Inje University Busan Paik Hospital, Busan
  - Korea University Ansan Hospital, Gyeonggi-do
  - Gachon University Gil Medical Center, Incheon
  - Hallym University Kangnam Sacred Heart Hospital, Seoul
- Spain (6):
  - Cs Algeciras Norte, Algeciras
  - Hosp. Gral. Univ. de Alicante, Alicante
  - Eap Sardenya, Barcelona
  - Cap Apenins - Montigala, Caldes Montbui Canovelles
  - Cap Canet de Mar, Canet de Mar
  - Hosp. Clinico San Carlos, Madrid
- Taiwan (6):
  - Kaohsiung Medical University Chung Ho Memorial Hospital, Kaohsiung City
  - Taipei Medical University Shuang Ho Hospital, New Taipei City
  - Taipei Medical University, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Tri-Service General Hospital, Taipei
  - Taipei Municipal Wanfang Hospital, Taipei
- The Adam Practice, Metropolitan Borough of Wirral, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson and Johnson is available at www.janssen.com/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency